CLINICAL TRIAL: NCT06486831
Title: The Effect of Stress Ball in Reducing Anxiety and Fear During Plastering Procedure in Extremity Fractures in Children Aged 6-12 Years
Brief Title: The Effect of Stress Ball in Reducing Anxiety and Fear in 6-12 Year Old Children
Acronym: TSA-2023-12759
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Zülbiye demir barbak, Lecturer, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: TSA-2023-12759
Record Dates: First submitted 2024-06-27; First posted 2024-07-05 (Actual); Last update posted 2024-07-05 (Actual); Status verified 2024-06

CONDITIONS: Plaster of Paris Injury to Skin
Keywords: Children; Plaster Intervention; Stress Ball; Anxiety; Fear; Trauma
MeSH Terms: conditions — Anxiety Disorders; Wounds and Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group (No Intervention): Routine Plaster intervention will be applied to the control group. No action will be taken.
- Experimental Group (Experimental): During the plaster intervention process, the experimental group will squeeze the stress ball.
  Interventions: Other: Squeeze the stress ball.

INTERVENTIONS:
Other: Squeeze the stress ball. — The child and parents will be taken to the procedure room for the casting procedure. The plastering process in children takes an average of 10-15 minutes. In the experimental group, the stress ball selected by the child will be started 1-2 minutes before the casting process and will be watched for an average of 10 minutes. If the procedure is prolonged, the time for squeezing and playing with the stress ball will be extended.
  Arms: Experimental Group

SUMMARY:
The aim of this study was to determine the effect of stress ball application on procedure-related anxiety and fear during plaster cast procedure in children aged 6-12 years.

DETAILED DESCRIPTION:
Children aged 6-12 years will be randomly divided into two groups: stress ball and control group. Interventions will be applied 1 time per day (2 sessions) for 2 days. Children in the experimental group will be given a stress ball during the plaster procedure and will be asked to squeeze it during the procedure. Children will be assessed before, during and after the intervention. Fear and anxiety related to the cast procedure will be assessed using the Children's Fear Scale, and the Children's Anxiety Scale - Statefulness Scale. In addition, children's heart rate, respiration, blood pressure and SPO2 will be measured.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 6 and 12 years (over 12 years old)
2. Absence of any physical and mental illness,
3. Not having taken analgesics in the last six hours
4. Hospitalization was for diagnostic or therapeutic purposes
5. The child and parents are comfortable speaking and understanding Turkish.

Exclusion Criteria:

1. Children hospitalized for surgery will not be included in the study.
2. Those who are outside the inclusion criteria will not be included in the study.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 116 (Estimated)
Dates: Start 2024-08-20 (Estimated); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-20 (Estimated)

PRIMARY OUTCOMES:
Patient Identification Form | baseline
  In this form, there are questions about the child's age, gender, weight, age of the mother and father, presence of long-term illness, previous hospitalization status and reason, previous surgery status, presence of medication on continuous use, analgesic intake in the last 6 hours.

SECONDARY OUTCOMES:
Children's Fear Scale (CFS) | baseline
  The CFS, which was first used in 2003, is a scale with proven validity and reliability developed to assess the child's fear/anxiety and its level. The scale includes five different facial expressions, with no fear/anxiety at one end and very intense fear/anxiety at the other end, and is evaluated on a 0-4 point scale. 0: no fear/anxiety, 4: extreme fear and anxiety.

OTHER OUTCOMES:
Child Anxiety Scale-Dispositional (CAS-D) | Baseline
  The CAS-D is shaped like a thermometer with a bulb at the bottom and horizontal lines with intervals going upwards. It is intended for children aged 4-10 years. The scale instructs children to "Imagine that all your anxious or angry feelings are at the bulb or bottom of the thermometer". Following the data collection, two members of the research team review and score the child's CAS-D scores. The score can range from 0 to 10.

CONTACTS AND LOCATIONS:
Overall Officials: Orhan DELİCE, 3, Study Chair — ERZURUM CITY HOSPİTAL

REFERENCES:
- [Result] Yurdakul Z, Esenay FI. Effects of two different ball types on pain and anxiety during venous blood draw in children: A randomized controlled study. J Pediatr Nurs. 2023 Sep-Oct;72:e201-e209. doi: 10.1016/j.pedn.2023.06.029. Epub 2023 Jul 5. PMID 37414624